CLINICAL TRIAL: NCT02855294
Title: The Effect of Oral Contraceptives on Dynamic Balance in Women
Brief Title: The Effect of Oral Contraceptives on Women Balance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 151
Record Dates: First submitted 2016-07-29; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Joint Stabilioty
Keywords: oral contraceptive pills; Joint stability
MeSH Terms: interventions — drospirenone; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral contraceptive pills users (Active Comparator): The participants received treatment for 6 consecutive cycles. Each treatment cycle consisted of 3 weeks of ring/pill treatment followed by a 1-week pill-free period. The women were randomized in a 1:1 ratio to receive the COC containing 30 μg of EE and 3mg of drospirenone (Yasmin; Schering AG, Berlin, Germany)
  Interventions: Drug: COC containing 30 μg of EE and 3mg of drospirenone
- control (No Intervention): no drugs

INTERVENTIONS:
Drug: COC containing 30 μg of EE and 3mg of drospirenone — treatment for 6 consecutive cycles. Each treatment cycle consisted of 3 weeks of pill treatment followed by a 1-week pill-free period.
  Other Names: Yasmin; Schering AG, Berlin, Germany
  Arms: Oral contraceptive pills users

SUMMARY:
1. Recording Data Sheet:

   All data and information of each woman in both groups (A & B) participated in this study were recorded in a recording data sheet (Appendix II).
2. Weight-Height scale:

   A valid and reliable weight -height scale, with a range of 1 to 150 kilograms weight, and 1 to 200 centimeters height was used to measure the relevant subject's data.
3. Siemens Immulite Immunoassay System:

   (Siemens Medical Solutions Diagnostics Immulite 1000,Los Angles, CA, 900-456900 U.S.A) to measure the serum Progesterone and Estradiol levels in both groups (A& B) using (TKE 21 Kit) for Estradiol and (TKPG 1 Kit) for Progesterone.
4. Biodex balance system:

Biodex Balance System (BBS), P.O. Box 702, Shirley, Ny 11967.It is an apparatus used to measure the dynamic balance. It utilizes dynamic multi axial platform. This platform allows approximately 20 degree inclination in 360 degree range and is interfaced with computer software. It measures the patient's ability to control the platform's angle of tilt, which is quantified as a variance from the center, as well as the degree of deflection over time at various stability levels as shown in (Fig. 6).

Stability levels allowed by the system ranged from one to eight. Stability level 8, allows the highest level of stability as it makes the platform to be the least tilted. On the other hand, stability level one represents the least level of stability and is more difficult for the subject to maintain stability on.

The test consists of recording the patient's ability to control the platform variance from a perfectly balanced position. A large variance is indicative of poor control and balance. Further definition is realized with the quantification of Anterior/ Posterior and Medial/Lateral responses.

DETAILED DESCRIPTION:
1. Recording Data Sheet:

   All data and information of each woman in both groups (A & B) participated in this study were recorded in a recording data sheet.
2. Weight-Height scale:

   A valid and reliable weight -height scale, with a range of 1 to 150 kilograms weight, and 1 to 200 centimeters height was used to measure the relevant subject's data.
3. Siemens Immulite Immunoassay System:

   (Siemens Medical Solutions Diagnostics Immulite 1000,Los Angles, CA, 900-456900 U.S.A) to measure the serum Progesterone and Estradiol levels in both groups (A& B) using (TKE 21 Kit) for Estradiol and (TKPG 1 Kit) for Progesterone.
4. Biodex balance system:

Biodex Balance System (BBS), P.O. Box 702, Shirley, Ny 11967.It is an apparatus used to measure the dynamic balance. It utilizes dynamic multi axial platform. This platform allows approximately 20 degree inclination in 360 degree range and is interfaced with computer software. It measures the patient's ability to control the platform's angle of tilt, which is quantified as a variance from the center, as well as the degree of deflection over time at various stability levels as shown in .

Stability levels allowed by the system ranged from one to eight. Stability level 8, allows the highest level of stability as it makes the platform to be the least tilted. On the other hand, stability level one represents the least level of stability and is more difficult for the subject to maintain stability on.

The test consists of recording the patient's ability to control the platform variance from a perfectly balanced position. A large variance is indicative of poor control and balance. Further definition is realized with the quantification of Anterior/ Posterior and Medial/Lateral responses.

The BBS Consists of the Following:

* Display Screen: Its height can be adjusted from 51cm to 68 cm above the platform. Display angle of the screen can be adjusted from vertical back up to 45º. Display viewing area: 122 mms x 92 mms. Display accuracy: ±1 degree of tilt.
* Support Handle Rails: Adjustable from 125 cm to 136.5 cm above the platform. The rails can be swung away from the platform if desired.
* Platform: Its height is 8 cm above floor, with a diameter of 21.5 cm. The platform has a grid which consists of two coordinates: X and Y. The platform X coordinate is marked in numbers from 1 to 21, whereas the platform Y coordinate is marked in letters from A to P, the platform is also marked in angles from 0º to 45º, for precise feet placement and documentation of the subject during the test procedures .
* Printer: Cannon Bubble-Jet Printer, centronics parallel interface.

Stability levels:

- Biodex balance system has been allowed for eight stability levels, which has been ranged from stability level (1) to stability level (8).which allows setting up of the test parameters.

Stability indices:

* The woman's ability to control the platform's angle of tilt measured by the system.The woman's performance wasnoted as a stability index.
* The stability index represents the variance of platform displacement in degrees from level. A high number is an indicative of a lot of motion, which indicates balance problem.
* The data regarding the balance of the tested woman were supplied to the system. These data includesantero-posterior stability index (APSI), medio-lateral stability index (MLSI) &overall stability index (OSI).
* On the upper most part of the surface of the platform appear angles from 0o to 95o with the lines which represents these angles. These lines would be used to measure foot angle.
* The smaller the amount of sway, the lower the numerical value of these indices.
* Over all stability index (OSI): Represents the woman's ability to control her balance in all directions.
* Anterior/Posterior stability index (APSI): Representsthe woman's ability to control her balance in front to back directions (sagittal plane).
* Medial/Lateral stability index (MLSI): Represents the woman's ability to control her balance from side to side directions(frontal plane).

III-Methods:

The evaluation procedures were explained in details for every woman in both groups (A&B) to increase her interest and co-operation.

Body Mass Index

The data of each woman in both groups were taken according to items of the recording data sheet then, the weight and height were measured and BMI was calculated according to the following equation BMI = Weight/Height (Kg/m2)

Blood sampling

Evening Blood sample was collected from each woman to limit the effect of hormone diurnal variations,For both groups samples have been collected at mid-luteal phase (20th to 23th days of the cycle), at Al-Madina Lab.

The sample was allowed to clot in water bath at room temperature.the serum was separated using a centrifuge at 4000 rmp for 15 min.Then using the TKE 21 and TKPG 1 Kits in a low temperature air conditioned room to measure serum Estradiol and Progesterone levels.

Biodex balance system:

The procedures were performed in dynamic balance lab at physical therapy faculty CairoUniversity.

Biodex Balance System used for assessment of the postural stability in female oral contraceptive users and non-users. The assessment was conducted for each woman individually.

The protocol of the work was explained to the woman before conducting this study.

A) Biodex balance system:

Operating the balance system:

* When the system is on, the first displayed screen showed the main menu. It allowed us to choose entering test or system utilities.
* Choosing to enter testing showed the next screen, which allowed for determining the test parameters as test duration and the stability levels were chosen as the initial stability level (8) and the end stability level (4).
* The next screen was used for centering process.
* The next screen was the stability test screen. The start key was pressed while on this screen to unlock the platform allowing the test to start. A cursor appeared during the test tracing the movement of the platform while the timer counting till the time of the test ends.
* The duration of test lasts for 20 seconds staring with stability level (8) and progressing the stability levels ending with stability level (4)
* The foot platform automatically returned to the locked position. At this point, the investigators printed the screen, including the numeric value of the APSI, MLSI and OSI.

Testing Protocol:

* Testing procedures was done at mid-luteal phase (20th to 23th days of the cycle). Each woman was received verbal explanation about the test steps.
* The woman was tested without footwear and with eyes opened.
* Two test trials was done before specific test condition for the purpose of instrument familiarity prior to data collection.
* A high stability level (stability level 8) and reduced test time (20 sec) was chosen to avoid falling.
* Each woman was asked to perform two trial tests and their mean was calculated.
* Each test started with the balance platform in the locked position and standing on its center.

Preparatory step: the parameters of each examined woman (weight, height and age) as well as, test duration and stability level of the platform of the BBS were typed to the software of the device as shown in Fig. (8). All woman were asked to stand on the platform of the BBS in an erect posture as possible and kept it all through the test duration (i.e. stand on both feet, chin in, shoulders were leveled, as well as, retracted , back was straight and knees were drawn backward). Hence, the support handle rails and display screen were adjusted according to the height of each examined woman.

Centering step: with the aim of positioning the center of gravity (COG) of the subject at the middle of her base of support between the two feet and recoding the women's feet position. Centering was achieved by asking each woman to stand on the platform of the BBS while grasping the support handle rails by both hands while the platform was locked . Formerly, the platform was unlocked at stability level 8, the display screen showed a circle with a central cursor. At that time, the subject was asked to achieve a central position on the platform by shifting her feet position until she was able to keep the cursor (which represents the center of platform) centered on the circle that appeared on the display screen and correspondingly the platform was kept easily leveled.

- Once centering was achieved and the cursor was in the center of the display screen, each woman was instructed to maintain her feet at that position constant until the end of test procedures. At that time, the platform was locked again to allow recording the feet angles and heel's coordinates from the platform grid. The heel's coordinates were determined by finding the location of the center of the back of each heel in relation to X and Y coordinates of the platform, while the feet angles were determined by finding a line on the platform parallel to the 2nd metatarsal bone of each foot. Then, the feet angles and heels coordinates for each womanwere entered to the software of the BBS

ELIGIBILITY:
Inclusion Criteria:

* All women in group (A) had takenthe oral contraceptive pill have done so routinely for the past three months.
* All women in group (B) had a normal menstrual cycle; use any other non-hormonal contraceptive method.
* Their body mass index did not exceed 30 Kg/m2.
* All women had a normal menstrual cycle of 25-32 days for the past 3 months.
* They can stand independently.

Exclusion Criteria:

* Respiratory or heart problems.
* Skeletal deformityorusing assistive devices.
* Visual and vestibular system affection.
* Cognition problems.
* Previous surgeries at their back and/or lower limbs.
* Genital and breast cancer and active liver disease.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
overall joint stability | 6 months after pill use
  A) Biodex balance system:
  Testing procedures was done at mid-luteal phase (20th to 23th days of the cycle). Each woman was received verbal explanation about the test steps.
  The woman was tested without footwear and with eyes opened. Two test trials was done before specific test condition for the purpose of instrument familiarity prior to data collection.
  A high stability level (stability level 8) and reduced test time (20 sec) was chosen to avoid falling.
  Each woman was asked to perform two trial tests and their mean was calculated. Each test started with the balance platform in the locked position and standing on its center.

SECONDARY OUTCOMES:
side effects | 6 months after pill use

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Maged AM, Salah E, Kamel AM, Hussein AM, Saad H, Meshaal H, Kamal WM. Effect of oral contraceptives on balance in women: A randomized controlled trial. Taiwan J Obstet Gynecol. 2017 Aug;56(4):463-466. doi: 10.1016/j.tjog.2017.02.003. PMID 28805601